CLINICAL TRIAL: NCT00839839
Title: Oocyte Cryopreservation in Assisted Reproduction
Brief Title: Egg Freezing Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Reproductive Associates (Other)
Responsible Party: Principal Investigator, Peter McGovern, MD, Principal Investigator, University Reproductive Associates
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 0120080226
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Infertility; Egg Freezing
Keywords: infertility; egg freezing; fertility preservation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oocyte Vitrification (Experimental)
  Interventions: Procedure: Oocyte Vitrification

INTERVENTIONS:
Procedure: Oocyte Vitrification — All oocytes retrieved will be vitrified (rapidly frozen) after egg retrieval. The oocytes will then be warmed on the same day and fertilized per standard IVF-ICSI. Resulting embryos will be transferred back to the patient as per protocol.

SUMMARY:
University Reproductive Associates is conducting a pilot study to study the technique of egg freezing. Your participation in this study will provide us with important information to allow us to offer this technology for women wishing to freeze their eggs before cancer treatments. Your participation will include a standard IVF cycle with your eggs being frozen for a brief period of time and then transferred back to you as usual. You will receive a significant reduction in your IVF cycle cost.

ELIGIBILITY:
Inclusion Criteria:

1. 10 women between the ages of 18-35 inclusive at time of signing Informed Consent Form.
2. In good general health off of current medications which may confound response to study medications.
3. Desire to seek pregnancy actively during the study period by IVF-ICSI.
4. A normal uterine cavity must have been confirmed by either hydrosonogram or hysteroscopy within two years of entering the study.
5. Ability to use the required medications.
6. Day 3 FSH level < 12 IU/ml

Exclusion Criteria:

1. Current pregnancy
2. Patients with significant anemia (Hemoglobin < 10 mg/dL).
3. Patients enrolled simultaneously into other investigative studies that would interfere with this research study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Biochemical Pregnancy | 1 year

SECONDARY OUTCOMES:
Recovery of viable oocytes | 1 year
incidence of fertilization | one year
embryo development (how many fertilized eggs undergo development to a more advanced stage) | 1 year
clinical pregnancy (fetal pole visible on transvaginal ultrasound) per cycle | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter G. McGovern, MD, Principal Investigator — UMDNJ-NJMS
Locations (1):
- University Reproductive Associates, Hasbrouck Heights, New Jersey, United States

REFERENCES:
- See also: Related Info — http://www.uranj.com